CLINICAL TRIAL: NCT06478888
Title: Association Between Cognitive Impairment and the Presence of Hearing Problems and Precarious Conditions
Acronym: PAC
Status: Not yet recruiting | Type: Observational
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP240443
Record Dates: First submitted 2024-06-03; First posted 2024-06-27 (Actual); Last update posted 2025-05-25 (Actual); Status verified 2025-05

CONDITIONS: Cognitive Dysfunction
Keywords: cognitive disorders; hearing impairment; precariousness
MeSH Terms: conditions — Cognitive Dysfunction; Hearing Loss

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
Cognitive disorders are extremely common. Alzheimer's disease is the most common cognitive disorder, with an estimated 800,000 to 1 million patients suffering from this neurodegenerative disorder in France. Cognitive disorders can also be observed in other common conditions such as Parkinson's disease and multiple sclerosis.

It has been shown that the presence of hearing impairment associated with cognitive disorders increases the latter. In addition, rare studies have shown that people in precarious situations are at greater risk of developing cognitive disorders early and rapidly, and consequently dementia.

The population of Seine Saint Denis (93) is known to be particularly affected by precariousness, which is why the investigators want to study its impact on patients with cognitive disorders associated with hearing impairment. These people need to be detected and supported in order to offer them a hearing aid that would improve or stabilize their cognitive state, or at least facilitate the rehabilitative management of their cognitive deficit.

DETAILED DESCRIPTION:
The aim of our project is to study the association between the severity of cognitive problems and precariousness in people with hearing problems

While the data on the link between deafness and cognitive impairment is well established (Manrique et al., 2023), the data published in PubMed is poor or even non-existent when the precariousness of the individuals is taken into account.

In 2018, DREES published the results of the Capacités, Aides et REssources des seniors (CARE) ménages, seniors section survey, carried out in 2015 and looking at the living conditions and difficulties encountered in the daily lives of people aged 60 or over living at home. It was reported that 4% of the 15.7 million people over 60 in the French population had hearing difficulties, i.e. they reported having great difficulty or not managing at all to hear a conversation in a silent room. These difficulties differed according to whether the subjects surveyed were men or women, and also according to their social category. People with a degree (≥ bac +3) are 60% less likely to have hearing problems than those without a degree. These differences are linked in particular to inequalities in occupational risks, lifestyle habits and access to healthcare throughout the life cycle, making the link between precariousness and deafness. They also have an impact on immediate access to corrective measures. The most common cause of hearing loss in adults is presbycusis (physiological alteration of hearing function associated with aging), which can generally be compensated for by wearing a hearing aid. Of these people, seven out of ten do not wear a hearing aid.

the investigators would therefore like to study prospectively, in patients seen at our Memory unit and presenting with a cognitive impairment defined by an MMSE score ≤ 24 (140 patients/year), whether the presence of a precarious situation associated with a hearing impairment is an aggravating factor in this cognitive impairment.

ELIGIBILITY:
Inclusion Criteria:

* Patient aged over 50
* Patient seen in our Memory unit for a cognitive complaint
* Patient with proven cognitive impairment (with or without hearing impairment) (MMSE ≤ 24)
* Patient not fitted with a hearing aid
* Patient with MMSE > 20 understands, reads and writes French well, if MMSE ≤ 20 needs to be accompanied by a relative.

Exclusion Criteria:

* Patient or relative refusing to take part in the study
* Absence of social security and AME
* Absence of cognitive disorders (MMSE>25)
* Cognitive disorder linked to a history of head trauma
* Patient under legal protection (guardianship, curatorship or safeguard of justice)
* Patients with a language barrier that may affect MMSE readings

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with cognitive problems associated with hearing impairment and/or precariousness
Sampling Method: Non-Probability Sample
Enrollment: 270 (Estimated)
Dates: Start 2025-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2027-11 (Estimated)

PRIMARY OUTCOMES:
MMSE score in subjects with or without hearing problems who are not fitted with hearing aids and in those in precarious and non-precarious situations | through study completion an average of 1 year
  to assess the association between the severity of cognitive impairment and the presence of precariousness and hearing impairment without hearing aids, in the population of Seine-Saint-Denis.

SECONDARY OUTCOMES:
association between the severity of cognitive disorders and the presence of precariousness and unaidable hearing disorders, as determined by neuropsychological tests with a hippocampal diagnostic orientation | through study completion an average of 1 year
  to assess the association between the severity of cognitive disorders and the presence of precariousness and unaidable hearing disorders, measured using neuropsychological tests other than the MMSE, in patients with cognitive disorders of hippocampal origin.
association between the severity of cognitive disorders and the presence of precariousness and unaidable hearing disorders, as determined by neuropsychological tests with a frontal diagnostic orientation | through study completion an average of 1 year
  to assess the association between the severity of cognitive disorders and the presence of precariousness and unaidable hearing disorders, measured using neuropsychological tests other than the MMSE, in patients with cognitive disorders of frontal origin.
association between the severity of cognitive disorders and the presence of precariousness and unaidable hearing disorders, as determined by neuropsychological tests with mixed hippocampal and frontal origin. | through study completion an average of 1 year
  to assess the association between the severity of cognitive disorders and the presence of precariousness and unaidable hearing disorders, measured using neuropsychological tests other than the MMSE,in patients with cognitive impairment of mixed hippocampal and frontal origin.
MMSE score in subjects with or without hearing problems who are not fitted with hearing aids and in those in precarious and non-precarious situations by distinguishing four groups of patients | through study completion an average of 1 year
  to assess the association between the severity of cognitive impairment and the presence of precariousness and hearing impairment without hearing aids
Other neuropsychological tests to assess cognitive functions such as praxis and visual-spatial perception | through study completion an average of 1 year
  To assess the association between precariousness, hearing problems without hearing aids and the severity of cognitive problems, measured using neuropsychological tests other than the MMSE, by distinguishing four groups of patients
Assess the quality of life of these patients | through study completion an average of 1 year
  Quality of life assessed by the SF-36 questionnaire

CONTACTS AND LOCATIONS:
Locations (1):
- Service de neurologie, Bobigny, France